CLINICAL TRIAL: NCT03968341
Title: Intraocular Concentrations Study (Aqueous Humor, Vitreous Humor) of Antibiotics After Local and/or Systemic Administration in Endophthalmitis
Brief Title: Study of Intraocular Concentrations (Aqueous Humor, Vitreous Humor) of Antibiotics After Local and/or Systemic Administration in Endophthalmitis
Acronym: CINEBIOPHTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Collaborators: Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINEBIOPHTA
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Endophthalmitis
Keywords: intraocular concentrations of antibiotics
MeSH Terms: conditions — Endophthalmitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intraocular antibiotic concentrations determination (Experimental): In the event that the patient develops unfavourably, the ophthalmologist include the patient in the trial.
  The patient is reviewed at 48 hours after the introduction of probabilistic antibiotic therapy for clinical reassessment and the return of microbiological test results. Following this inclusion, the new samples will be taken when the patient passes through the operating room for the treatment of his pathology as part of the care. Ophthalmologists may have to adapt the patient's management (i.e. adjustment of antibiotic therapy) as part of their usual care routine. An anterior chamber puncture and a vitrectomy are performed. Eye fluids collected as part of the treatment are sent for analysis.
  Interventions: Other: Pharmacokinetic and pharmacodynamic study of antibiotics used in severe endophthalmitis from samples taken from treated patients

INTERVENTIONS:
Other: Pharmacokinetic and pharmacodynamic study of antibiotics used in severe endophthalmitis from samples taken from treated patients — A 5mL dry tube will be taken by puncture of the humeral vein like a conventional blood test. This tube is not usually collected unless specifically requested by the ophthalmologist. This sample will be sent quickly (within two hours) to the CHNO Medical Biology Laboratory for centrifugation, serum separation and storage at -80°C.
  Samples stored at -80°C will be sent weekly to the Microbiology and Anti-infectives Laboratory at Hospital Paris Saint-Joseph, with the dosage request form duly completed with the usual information.

SUMMARY:
Endophthalmitis is an intraocular inflammation due to a serious infection of bacterial, fungal or parasitic origin, involving visual prognosis if it is not treated in time and correctly. Despite the eye isolation from the rest of the body, germs can enter the eye either exogenously, during open globe surgery, following perforating eye trauma, or following anti-VEGF antibodies intravitreal injection, or other drugs such as corticosteroids for example, or by endogenous route, haematogenic as part of sepsis, usually during immunodepression. Post-operative endophthalmitis is the most feared complication following any endo-ocular surgery. It can be acute, occurring within 6 weeks post-operatively or delayed as after poor healing, or on a glaucoma filtration bubble. Endophthalmitis after cataract surgery is a complication with a low incidence of (0.030 to 0.047%) but which, due to interventions number carried out (830,000 in 2016, in France), appears significant. There are factors that favour endophtalmitis occurrence such as a vitreous exit from eyeball during surgical procedure, poor scar coaptation, premature removal of sutures, etc... They condition emergency care. Early diagnosis and appropriate treatment are essential for safeguarding the eye and its function. Therefore, therapeutic management requires endo-ocular sampling in front of any suspicion of endophtalmitis, to be done before any treatment, to carry out microbiological analysis (direct examination on slide, culture, universal and/or targeted PCR, antibiotic susceptibility test). Vitreous puncture is more contributive than anterior chamber puncture, underlining need for these two samples to identify the responsible germ. Once samples have been taken, a broad-spectrum antibiotic therapy introduction must be performed intra-vitreously combined with systemic and local administration. Intravitreal injections allow treatment to be provided at effective concentrations directly at the infection site. On the other hand, toxic risks must be taken into account, especially since the protocol may require multiple intravitreal injections.

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 18 years old
* Francophone
* Patients referred to emergencies by an ophthalmologist or doctor, or patients already hospitalized, with a unfavourable course 48 hours after introduction of broad spectrum probabilistic antibiotic therapy for the following situations:

  * Cataract surgery
  * Vitreoretinal surgery
  * Intravitreal injection [anti-VEGF for the treatment of AMD, dexamethasone (Ozurdex®) for the treatment of cystoid macular edema]
  * Physical signs presence of intraocular inflammation (Tyndall, hypopyon, cyclic membrane, hyalite)
  * Presence of functional signs (Decreased Visual Acuity)
* Patients for whom a management re-evaluation is essential with obligation of new intraocular samples.
* Patient affiliated to social security or, failing that, to another health insurance system

Exclusion Criteria:

* Patient under guardianship or curators
* Patient deprived of liberty
* Participation refusal in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2023-12-08 (Estimated)

PRIMARY OUTCOMES:
Determination of the concentrations of the various antibiotics in the media tested (aqueous and vitreous humours) | 48 hours
  Determination of the concentrations of the various antibiotics in the media tested (aqueous and vitreous humours) by liquid chromatography coupled with a high-resolution mass spectrometer (HPLC-HRMS).

SECONDARY OUTCOMES:
Number of aqueous or vitreous humor samples collected by puncture from treated patients that can be used analytically | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: François COUDORE, Professor, Study Director — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

REFERENCES:
- [Result] Du DT, Wagoner A, Barone SB, Zinderman CE, Kelman JA, MaCurdy TE, Forshee RA, Worrall CM, Izurieta HS. Incidence of endophthalmitis after corneal transplant or cataract surgery in a medicare population. Ophthalmology. 2014 Jan;121(1):290-298. doi: 10.1016/j.ophtha.2013.07.016. Epub 2013 Aug 29. PMID 23993357
- [Result] Clarke B, Williamson TH, Gini G, Gupta B. Management of bacterial postoperative endophthalmitis and the role of vitrectomy. Surv Ophthalmol. 2018 Sep-Oct;63(5):677-693. doi: 10.1016/j.survophthal.2018.02.003. Epub 2018 Feb 15. PMID 29453989
- [Result] Goldschmidt P, Bensaid P, Semoun O, Chaumeil C. [Rational approach for the treatment of postoperative endophthalmitis in impoverished populations]. J Fr Ophtalmol. 2013 Mar;36(3):261-7. doi: 10.1016/j.jfo.2012.08.002. Epub 2013 Feb 11. French. PMID 23410853
- [Result] Kumar A, Sridhar MS, Dada T, Tewari HK, Gupta SK. Intravitreal pefloxacin therapy in postoperative endophthalmitis. Clin Exp Ophthalmol. 2000 Feb;28(1):38-40. doi: 10.1046/j.1442-9071.2000.00256.x. PMID 11345344
- [Result] Khera M, Pathengay A, Jindal A, Jalali S, Mathai A, Pappuru RR, Relhan N, Das T, Sharma S, Flynn HW. Vancomycin-resistant Gram-positive bacterial endophthalmitis: epidemiology, treatment options, and outcomes. J Ophthalmic Inflamm Infect. 2013 Apr 22;3(1):46. doi: 10.1186/1869-5760-3-46. PMID 23607574
- [Result] Chiquet C, Labetoulle M. [Fluoroquinolones in ophthalmology: indications and current use]. J Fr Ophtalmol. 2008 Oct;31(8):803-8. doi: 10.1016/s0181-5512(08)74403-6. French. PMID 19107048
- [Result] Adenis JP, Mounier M, Salomon JL, Denis F. Human vitreous penetration of imipenem. Eur J Ophthalmol. 1994 Apr-Jun;4(2):115-7. doi: 10.1177/112067219400400207. PMID 7950335
- [Result] Bowen RC, Zhou AX, Bondalapati S, Lawyer TW, Snow KB, Evans PR, Bardsley T, McFarland M, Kliethermes M, Shi D, Mamalis CA, Greene T, Rudnisky CJ, Ambati BK. Comparative analysis of the safety and efficacy of intracameral cefuroxime, moxifloxacin and vancomycin at the end of cataract surgery: a meta-analysis. Br J Ophthalmol. 2018 Sep;102(9):1268-1276. doi: 10.1136/bjophthalmol-2017-311051. Epub 2018 Jan 11. PMID 29326317
- [Result] Cornut PL, Chiquet C. [Intravitreal injection of antibiotics in endophthalmitis]. J Fr Ophtalmol. 2008 Oct;31(8):815-23. doi: 10.1016/s0181-5512(08)74405-x. French. PMID 19107050
- [Result] Gan IM, van Dissel JT, Beekhuis WH, Swart W, van Meurs JC. Intravitreal vancomycin and gentamicin concentrations in patients with postoperative endophthalmitis. Br J Ophthalmol. 2001 Nov;85(11):1289-93. doi: 10.1136/bjo.85.11.1289. PMID 11673290
- [Result] Thompson AM. Ocular toxicity of fluoroquinolones. Clin Exp Ophthalmol. 2007 Aug;35(6):566-77. doi: 10.1111/j.1442-9071.2007.01552.x. PMID 17760640